CLINICAL TRIAL: NCT02549391
Title: Phase 3 Study of KHK7580 (A Randomized, Double-Blind, Intra-Subject Dose-Adjustment, Parallel-Group Study of KHK7580 and Cinacalcet Hydrochloride in Subjects With Secondary Hyperparathyroidism Receiving Hemodialysis)
Brief Title: Phase 3 Study of KHK7580
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7580-010
Record Dates: First submitted 2015-09-09; First posted 2015-09-15 (Estimated); Last update posted 2017-03-24 (Actual); Status verified 2017-03

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary | interventions — Cinacalcet

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KHK7580 (Experimental)
  Interventions: Drug: KHK7580
- KRN1493 (Active Comparator)
  Interventions: Drug: KRN1493

INTERVENTIONS:
Drug: KHK7580 — Oral administration
  Arms: KHK7580
Drug: KRN1493 — Oral administration
  Other Names: cinacalcet hydrochloride
  Arms: KRN1493

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of KHK7580 orally administered once daily for 30 weeks in subjects with secondary hyperparathyroidism (SHPT) receiving hemodialysis in a randomized, double-blind, intra-subject dose-adjustment, parallel-group design with cinacalcet hydrochloride as an active control.

ELIGIBILITY:
Inclusion Criteria:

* Personally submitted written voluntary informed consent to participate in the study
* Stable chronic renal disease treated with hemodialysis 3 times weekly for at least 12 weeks before screening
* Mean intact PTH level of > 240 pg/ml at screening, at 2 weeks and 1 week before the start of study treatment

Exclusion Criteria:

* Treatment with cinacalcet hydrochloride within 2 weeks before screening;
* Change in dose or dosing regimen of an activated vitamin D drug or its derivative, phosphate binder, or calcium preparation within 2 weeks before screening; or start of treatment with such drugs within 2 weeks before screening;
* Parathyroidectomy and/or parathyroid intervention within 24 weeks before screening;
* Severe heart disease;
* Severe hepatic dysfunction;
* Uncontrolled hypertension and/or diabetes;
* Treatment with an investigational product (drug or medical device) in a clinical study or any study equivalent to clinical study within 12 weeks before screening;
* Primary hyperparathyroidism;
* Other conditions unfit for participation in this study at the discretion of the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 634 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects in the evaluation period achieving a mean intact parathyroid hormone (PTH) level of ≥ 60 pg/mL and ≤ 240 pg/mL | Weeks 28-30

SECONDARY OUTCOMES:
Percentage of subjects in the evaluation period achieving a mean percent decrease in intact PTH level of ≥ 30% (percent change ≤ -30%) from baseline | Weeks 28-30
Mean percent change in the evaluation period in intact PTH level from baseline | Weeks 28-30

CONTACTS AND LOCATIONS:
Locations (1):
- For additional information regarding investigative sites for this trial, contact Kyowa Hakko Kirin, Tokyo, Japan

REFERENCES:
- [Derived] Tokumoto M, Tokunaga S, Asada S, Endo Y, Kurita N, Fukagawa M, Akizawa T. Predictive factors requiring high-dose evocalcet in hemodialysis patients with secondary hyperparathyroidism. PLoS One. 2022 Dec 13;17(12):e0279078. doi: 10.1371/journal.pone.0279078. eCollection 2022. PMID 36512619
- [Derived] Shigematsu T, Asada S, Endo Y, Kawata T, Fukagawa M, Akizawa T. Evocalcet with vitamin D receptor activator treatment for secondary hyperparathyroidism. PLoS One. 2022 Feb 17;17(2):e0262829. doi: 10.1371/journal.pone.0262829. eCollection 2022. PMID 35176038